CLINICAL TRIAL: NCT00513734
Title: Randomised Trial Comparing the Efficacy of Ocular Lubricant (Lacrilube) and Polyacrylamide Hydrogel Dressing (Geliperm) for the Prevention of Exposure Keratopathy in the Critically Ill
Brief Title: A Comparison of Hydrogel Dressings and Ocular Lubricants in the Prevention on Corneal Damage in the Critically Ill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 003171
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Keratitis
Keywords: keratopathy; exposure; intensive care; eye; ulcer; Corneal
MeSH Terms: conditions — Keratitis; Ulcer | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Geliperm Hydrogel Dressing
  Interventions: Other: Hydrogel dressing
- 2 (Active Comparator): Lacrilube ointment
  Interventions: Other: Lacrilube ointment

INTERVENTIONS:
Other: Hydrogel dressing — 3x3cm hydrogel dressing over closed eye
  Arms: 1
Other: Lacrilube ointment — lubricant put into eye (inferior formix)
  Arms: 2

SUMMARY:
Corneal damage in critically ill patients is common. There are currently two popular methods of treatment in the UK; hydrogel dressings and lubricating ointment. We propose to randomise patients to have a different treatment for each eye and see which one is more effective.

DETAILED DESCRIPTION:
Microbial keratitis, particularly pseudomonas-related, has been widely reported amongst Intensive therapy unit (ITU) patients and the need for effective eye care in ITU has been recognised for some time. We compare two popular methods of eye care; a hydrogel dressing and lacrilube ointment. Each recruited patient had each eye randomised to different treatments. Daily ophthalmology ward rounds were undertaken to identify any corneal exposure keratopathy. Patients were removed from the trial if one eye developed significant exposure needing treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Intensive care and expected to stay for more than 2 days

Exclusion Criteria:

* Primary orbital injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-09; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Development of clinically significant corneal exposure | throughout length of admission to ITU

CONTACTS AND LOCATIONS:
Overall Officials: Marie Healy, FRCA, Study Director — Lead Clinicain, Dept. of Intensive Care Medicine, Royal London Hospital, London E1 1BB